CLINICAL TRIAL: NCT05092568
Title: Comparison of General Characteristics of Patients Diagnosed COVID-19 Positive Followed In Service
Brief Title: Comparison of General Characteristics of Patients Diagnosed COVID-19 (Coronavirus )Positive Followed In Service
Acronym: COVID-19
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Saglik Bilimleri Universitesi (Other)
Responsible Party: Principal Investigator, Sevim Özge Özdemir, Doctor, Saglik Bilimleri Universitesi
Other Study IDs: COVID-19
Record Dates: First submitted 2021-10-22; First posted 2021-10-25 (Actual); Last update posted 2022-05-06 (Actual); Status verified 2022-05

CONDITIONS: Coronavirus Disease 2019; Vaccinia; Symptoms and Signs
Keywords: covid 19,; vaccine; covid pregnancy vaccine
MeSH Terms: conditions — COVID-19; Vaccinia; Signs and Symptoms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- covid pregnancy: Pregnant patients with positive polymerase chain reaction assay COVID-19 test results, who were followed up and treated in the pandemic service of Başakşehir Çam and Sakura City Hospital.

SUMMARY:
comparison of general characteristics of patients diagnosed COVID-19 positive followed In service

DETAILED DESCRIPTION:
After the explanation about the study is made, informed consent form will be obtained from the pregnant women who were hospitalized in the pandemic gynecology service (D block 10th floor pandemic obstetrics service) due to COVID-19 and who agreed to participate in the study. In our study, the clinical status of pregnant patients with COVID-19 positive test results, who were followed up and treated in the pandemic service in Basaksehir City Hospital, will be obtained by asking the patient about the symptoms and vaccination status in the patient follow-up form prepared in advance. Laboratory findings and imaging results ( CT/ anteroposterior X-ray) will be obtained from the recorded data.

ELIGIBILITY:
Inclusion Criteria: Pregnant patients positive COVID-19 test results followed up and treated in the pandemic service of Çam and Sakura City Hospital.

Exclusion Criteria: no exclusion criteria

-

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Pregnant patients with positive COVID-19 test results, who were followed up and treated in the pandemic service of Çam and Sakura City Hospital.
Sampling Method: Probability Sample
Enrollment: 45 (Estimated)
Dates: Start 2022-05-05 (Actual); Primary Completion 2022-07-15 (Estimated); Study Completion 2022-07-15 (Estimated)

PRIMARY OUTCOMES:
Number of Participants | Two months
  Number of Participants diagnosed of polymerase chain reaction assay Positive COVID-19 followed İn service
Number of vaccinated participants | Two months
  Vaccinated patients who were followed up in the service due to COVID-19
Number of non-vaccinated Participants | Two months
  non-vaccinated patients who were followed up in the service due to COVID-19
rate of non-vaccinated -vaccinated Participants | Two months
  rate of non-vaccinated- vaccinated Participants who were followed up in the service due to COVID-19
rate of covid symptoms | Two months
  rate of covid common symptoms (cough, fever, shortness of breath ,sore throat ) in vaccinated and unvaccinated patients
rate of inflammatory parameters | Two months
  rate of lymphocyte and albumin levels , C-reactive protein (CRP), D-dimer, Ferritin, lactate dehydrogenase(LDH), neutrophil lymphocyte ratio (NLR), platelet lymphocyte ratio (PLR) and C-reactive protein albumin ratio (CAR) levels in vaccinated and unvaccinated patients

CONTACTS AND LOCATIONS:
Overall Officials: Ozge Ozdemir, Principal Investigator — Saglik Bilimleri Universitesi
Locations (1):
- Department of Obstetrics and Gynecology, Maternal-Fetal Medicine Unit, Başakşehir City Hospital, Hamidiye School of Medicine, University of Health Sciences,, Başaksehir, Istanbul, Turkey (Türkiye)